CLINICAL TRIAL: NCT04394286
Title: An Open-Label, Multinational, Phase 1/2 Study of the Safety and Dose Escalation of SHP648, an Adeno-Associated Virus Serotype 8 (AAV8) Vector Expressing FIX Padua in Hemophilia B Subjects
Brief Title: A Phase 1/2 Study of SHP648, an Adeno-Associated Viral Vector for Gene Transfer in Hemophilia B Subjects
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Takeda has decided to not further develop the SHP648 (TAK-748) program. No subjects have been dosed with SHP648. The decision to terminate study SHP648-101 is not due to any safety concerns.
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SHP648-101; 2018-004024-11 (EudraCT Number)
Record Dates: First submitted 2020-05-15; First posted 2020-05-19 (Actual); Results first posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-04

CONDITIONS: Hemophilia B
MeSH Terms: conditions — Hemophilia B

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Cohort 1 participants will receive a single intravenous (IV) infusion of SHP648 on the day of dosing (Day 0).
  Interventions: Genetic: SHP648
- Cohort 2 (Experimental): Cohort 2 participants will receive a single IV infusion of SHP648 at a 2 to 3-fold escalation of Cohort 1 on the day of dosing (Day 0).
  Interventions: Genetic: SHP648
- Cohort 3 (Experimental): Cohort 3 participants will receive a single IV infusion of SHP648 at a 2 to 3-fold escalation of Cohort 2 on the day of dosing (Day 0).
  Interventions: Genetic: SHP648

INTERVENTIONS:
Genetic: SHP648 — Participants will receive a single IV infusion of SHP648 in Cohort 1, 2, 3 on Day 0.
  Other Names: TAK748; AAV8.ss-3xCRM8-TTR-FIX_R338Lopt

SUMMARY:
The purpose of this study is to evaluate the safety and dose escalation of SHP648 an adeno-associated viral vector for gene transfer in hemophilia B participants.

DETAILED DESCRIPTION:
This study will consists of 3 dose cohorts with 2-7 participants in each of the three ascending dose cohorts. Initially 2 participants will be dosed in Cohort 1, followed by dosing of up to 5 additional participants if the cohort is expanded. Participants in cohort 2 and 3 will receive 2-fold or 3-fold dose escalation to their respective preceding cohort doses if required.

ELIGIBILITY:
Inclusion Criteria:

* Male, aged 18 to 75 years at the time of screening.
* Established severe or moderately severe hemophilia B (plasma FIX activity lesser than or equal to [<=] 2 percent (%) measured following greater than or equal to [>=] 5 half-lives of most recent exposure to exogenous FIX) and either >= 3 hemorrhages per year requiring treatment with exogenous FIX or use of prophylactic therapy.
* History of greater than (>) 50 exposure days to exogenously administered FIX concentrates or cryoprecipitates.
* Sexually active men must agree to use barrier contraception (combination of a condom and spermicide) or limit sexual intercourse to post-menopausal, surgically sterilized, or contraception-practicing partners for a minimum of 6 months after administration of SHP648, or until SHP648 genomes are no longer detected in the semen (whichever is sooner).
* Signed informed consent.

Exclusion Criteria:

* Bleeding disorder(s) other than hemophilia B.
* Documented laboratory evidence of having developed inhibitors (>= 0.6 Bethesda Units [BU] on any single test) to FIX proteins at any time.
* Documented prior allergic reaction to any FIX product.
* Anti-AAV8 neutralizing antibody titer >= 1:5.
* Known hypersensitivity to prednisolone or prednisone, or to any of the excipients.
* Having a disease in which treatment with prednisolone or prednisone is not tolerated (including, but not limited to osteoporosis with vertebral fractures, severe labile hypertension, and brittle diabetes).
* Evidence of markers of potential underlying risk for autoimmune mediated hepatic disease:

  * Anti-smooth muscle antibody (ASMA) titer >= 1:40. Values of 1:31 to 1:39 will be flagged as possibly abnormal and the Investigator and Medical Monitor will evaluate the participant for eligibility
  * Elevated anti-liver-kidney microsomal antibody type 1 (LKM1) titers
  * Total Immunoglobulin G (IgG) > 1.5x upper limit of normal (ULN)
  * Antinuclear antibody (ANA) titer > 1:320 OR ANA titer > 1:80 if demonstrated concurrently with alanine aminotransferase (ALT) that is > ULN
* Active Hepatitis C: as indicated by detectable hepatitis C virus ribonucleic acid (HCV RNA) by polymerase chain reaction (PCR).
* Hepatitis B: If surface hepatitis B virus (HBV) antigen is positive.
* Receiving chronic systemic antiviral and/or interferon therapy within 4 weeks prior to enrollment.
* Clinically significant infections (e.g., systemic fungal infections) requiring systemic treatment.
* Known immune disorder (including myeloma and lymphoma).
* Concurrent chemotherapy or biological therapy for treatment of neoplastic disease or other disorders.
* An absolute neutrophil count lesser than < 1000 cells per cubic millimetre (cells/mm^3).
* Markers of hepatic inflammation or cirrhosis as evidenced by 1 or more of the following:

  * Platelet count < 150,000/microliter (μL)
  * Albumin <= 3.5 gram per deciliter (g/dL)
  * Total bilirubin > 1.5x ULN and direct bilirubin >= 0.5 milligram per deciliter (mg/dL)
  * ALT or Aspartate aminotransferase (AST) > 1.0x ULN
  * Alkaline phosphatase > 2.0x ULN
  * History of liver biopsy or imaging indicating moderate or severe fibrosis (Metavir staging of F2 or greater)
  * History of ascites, varices, variceal hemorrhage, or hepatic encephalopathy
  * FibroSURE Score >= 0.4
  * Prothrombin time international normalized ratio (INR) >= 1.4
* Serum creatinine > 1.5 mg/dL.
* Human immunodeficiency virus (HIV) if cluster of differentiation 4 (CD4)+ cell count <= 200 mm^3 and/or viral load > 20 copies per milliliter (copies/mL).
* Urine protein > 30 mg/dL.
* Body mass index > 38.
* Orthopedic or other major surgery planned within 6 months after enrollment.
* Acute or chronic disease that, in the opinion of the Investigator, would adversely affect participant safety or compliance or interpretation of study results.
* Received an AAV vector previously or any other gene transfer agent in the previous 12 months prior to Study Day 0.
* Significant cardiovascular disease (such as New York Heart Association Class III or IV cardiac disease, congestive heart failure, myocardial infarction within the previous 6 months, unstable arrhythmias, or unstable angina) or significant pulmonary disease (including obstructive pulmonary disease).
* History of arterial or venous thrombosis / thromboembolism, or a known pro-thrombotic condition.
* Recent history of psychiatric illness or cognitive dysfunction (including drug or alcohol abuse) that, in the opinion of the Investigator, is likely to impair participants ability to comply with protocol mandated procedures.
* Participation in another study involved with an investigational agent.
* Participant is family member or employee of the Investigator.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-05-13 (Actual); Primary Completion 2021-05-03 (Actual); Study Completion 2021-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Shire
Locations (2):
- Hospital Universitario Virgen de la Arrixaca, El Palmar, Spain
- Ege University Medical Faculty, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data from this particular study will not be shared as there is a reasonable likelihood that individual patients could be re-identified (due to the limited number of study participants/study sites)

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f6b5fe84db2bf003ab47acb

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study was terminated by the Sponsor. Only 2 participants were screened and signed informed consent but none received any treatment during this study. No participants were evaluated, and no data was collected to be reported here, in order to protect and maintain participant's privacy/confidentiality.
Groups:
- Cohort 1: SHP648: Cohort 1 participants were planned to receive a single intravenous (IV) infusion of SHP648 at dose 4.0*10^11 vector genome (vg) per kilogram (kg) body weight (BW) on the day of dosing (Day 0).
- Cohort 2: SHP648: Cohort 2 participants were planned to receive a single IV infusion of SHP648 at dose 8.0*10^11 vg/kg BW or 1.2*10^12 vg/kg BW on the day of dosing (Day 0). The dosing of Cohort 2 was to be decided upon evaluation of Cohort 1 data and recommendation from an external Data Monitoring Committee.
- Cohort 3: SHP648: Cohort 3 participants were planned to receive a single IV infusion of SHP648 at dose 1.6*10^12 vg/kg BW or 2.4*10^12 vg/kg BW or 3.6*10^12 vg/kg BW on the day of dosing (Day 0). The dosing of Cohort 3 was to be decided upon evaluation of Cohort 2 data and recommendation from an external Data Monitoring Committee.
Period: Overall Study
Arm/Group | Cohort 1: SHP648 | Cohort 2: SHP648 | Cohort 3: SHP648
Started | 0 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated by the Sponsor. Only 2 participants were screened and signed informed consent but none received any treatment during this study. No participants were evaluated, and no data was collected to be reported here, in order to protect and maintain participant's privacy/confidentiality.
Groups:
- Cohort 1: SHP648: Cohort 1 participants were planned to receive a single IV infusion of SHP648 at dose 4.0*10^11 vg/kg BW on the day of dosing (Day 0).
- Total: Total of all reporting groups
Arm/Group | Cohort 1: SHP648 | Cohort 2: SHP648 | Cohort 3: SHP648 | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Continuous [unit: years]
Sex: Female, Male [unit: participants]
Race/Ethnicity, Customized [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With SHP648 Related Serious and Non- Serious Adverse Events (AEs)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and that did not necessarily have a causal relationship with this investigational product (IP) or medicinal product. A Serious adverse event (SAE) was an AE resulting in any of the following outcomes: death; Life-threatening event; required or prolonged inpatient hospitalization; persistent or significant disability/incapacity; congenital anomaly.
Time Frame: From study start date to Month 12
Population: as for baseline characteristics
Arm/Group | Cohort 1: SHP648 | Cohort 2: SHP648 | Cohort 3: SHP648
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Plasma Factor IX (FIX) Levels Before and After SHP648 Infusion
Description: Plasma FIX levels before and after SHP648 infusion were planned to be reported.
Time Frame: From study start date to Month 12
Population: as for baseline characteristics
Arm/Group | Cohort 1: SHP648 | Cohort 2: SHP648 | Cohort 3: SHP648
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Annualized Bleed Rate (ABR) Before and After SHP648 Infusion
Description: ABR was to be assessed based upon each individual bleeding episode. A bleed episode was defined as subjective (example, pain consistent with a joint bleed) or objective evidence of bleeding which may or may not require treatment with FIX. ABR before and after SHP648 administration was planned to be reported.
Time Frame: From study start date to Month 12
Population: as for baseline characteristics
Arm/Group | Cohort 1: SHP648 | Cohort 2: SHP648 | Cohort 3: SHP648
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Number of Participants With Positive Binding Antibody Titers to Adeno-Associated Virus (AAV8)
Description: Number of participants with positive binding antibodies titers to AAV8 was planned to be reported.
Time Frame: From study start date to Month 12
Population: as for baseline characteristics
Arm/Group | Cohort 1: SHP648 | Cohort 2: SHP648 | Cohort 3: SHP648
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Number of Participants With Positive Neutralizing Antibody Titers to AAV8
Description: Number of participants with positive neutralizing antibodies to AAV8 was planned to be reported.
Time Frame: From study start date to Month 12
Population: as for baseline characteristics
Arm/Group | Cohort 1: SHP648 | Cohort 2: SHP648 | Cohort 3: SHP648
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With T-cell Response to AAV8
Description: Number of participants with T-cell response to AAV8 was planned to be reported.
Time Frame: From study start date to Month 12
Population: as for baseline characteristics
Arm/Group | Cohort 1: SHP648 | Cohort 2: SHP648 | Cohort 3: SHP648
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With T-cell Response to FIX Transgene Products
Description: Number of participants with T-cell response to FIX transgene products was planned to be reported.
Time Frame: From study start date to Month 12
Population: as for baseline characteristics
Arm/Group | Cohort 1: SHP648 | Cohort 2: SHP648 | Cohort 3: SHP648
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Duration of SHP648 Genomes Present in Bodily Fluids
Description: Duration of SHP648 genomes present in bodily fluids such as serum, blood, saliva, urine, stool, and semen was planned to be reported.
Time Frame: From study start date to Month 12
Population: as for baseline characteristics
Arm/Group | Cohort 1: SHP648 | Cohort 2: SHP648 | Cohort 3: SHP648
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Percent Change in Consumption of FIX Before and After Gene Transfer
Description: Percent change in consumption of exogenous FIX before and after gene transfer was planned to be reported.
Time Frame: From study start date to Month 12
Population: as for baseline characteristics
Arm/Group | Cohort 1: SHP648 | Cohort 2: SHP648 | Cohort 3: SHP648
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From study start date to Month 12
Description: The study was terminated by the Sponsor. Only 2 participants were screened and signed informed consent but none received any treatment during this study. No participants were evaluated, and no data was collected to be reported here, in order to protect and maintain participant's privacy/confidentiality.
Arm/Group | Cohort 1: SHP648 | Cohort 2: SHP648 | Cohort 3: SHP648
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study was terminated by the Sponsor. Only 2 participants were screened and signed informed consent but none received any treatment during this study. No participants were evaluated, and no data was collected to be reported here, in order to protect and maintain participant's privacy/confidentiality.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (1):
  • Study Protocol (2020-02-21): https://cdn.clinicaltrials.gov/large-docs/86/NCT04394286/Prot_002.pdf